CLINICAL TRIAL: NCT05089942
Title: Efficacy and Safety of Recombinant Human Insulin Patch ZJSRM2021 in Healthy and Diabetic Patients
Brief Title: Efficacy and Safety of Recombinant Human Insulin Patch ZJSRM2021
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao Ye, MD, Doctor, Zhejiang Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZJSRM2021
Record Dates: First submitted 2021-10-20; First posted 2021-10-22 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: type1diabetes; Type2 Diabetes
Keywords: insulin patch; type 1 diabetes mellitus; type 2 diabetes mellitus; safety; efficacy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant Human Insulin Patch ZJSRM2021 (Experimental): health subjects or diabetic patients receive recombinant human insulin patch ZJSRM2021
  Interventions: Drug: Recombinant Human Insulin Patch ZJSRM2021
- Placebo (Placebo Comparator): health subjects receive patch
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Recombinant Human Insulin Patch ZJSRM2021 — health subjects receive recombinant human insulin patch ZJSRM2021，diabetic patients receive recombinant human insulin patch ZJSRM2021（low-dosage or high dosage）
  Arms: Recombinant Human Insulin Patch ZJSRM2021
Drug: Placebo — health subjects receive placebo patch
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the efficacy，safety， and tolerability of the recombinant human insulin patch ZJSRM2021 in healthy subjects, type 1diabetes mellitus and type 2diabetes mellitus patients

ELIGIBILITY:
Inclusion Criteria:

* Type 1or type 2 diabetes Body mass index：19~35kg/m2（include） HbA1c≤11.0% Diabetic duration of T1DM was ≥1 year, and the subjects received insulin injections during the past year .Metformin and glycosidase inhibitors were also allowed.

Newly diagnosed T2DM or metformin-only, and the drug dose remained stable for ≥30 days. Or T2DM patients withdrawed drug ≥30 days of drug after diagnosis.

Exclusion Criteria:

* other type diabetes Use of other oral antidiabetics drugs within the 1 months prior to screening. With a history of malignant tumor. With acute or chronic infection. With evidence of major active psychiatric disorders. Drug abuse or alcohol abuse. Drunk too much tea or coffee(more than 2000ml per day). History of any drug allergies. Anti-insulin antibody positive. Participated in clinical trials within 3 months prior to signing the informed consent.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Recombinant Human Insulin Patch ZJSRM2021 | maximum 1 years
  the glucose and insulin level after receiving Recombinant Human Insulin Patch ZJSRM2021

SECONDARY OUTCOMES:
Incidence of adverse event of Recombinant Human Insulin Patch ZJSRM2021 | maximum 1 years
  Any adverse event(such as tachycardia, hypertension, hypoglycemia，coma) of Recombinant Human Insulin Patch ZJSRM2021
Skin irritation assessment and pain assessment of Recombinant Human Insulin Patch ZJSRM2021 | maximum 1 years
  Skin irritation assessment（Score range from 0：no irritation to 7：Intense stimulation such as blisters exceeds the patch coverage) after receiving Recombinant Human Insulin Patch ZJSRM2021
Pain assessment of Recombinant Human Insulin Patch ZJSRM2021 | maximum 1 years
  Pain assessment（Visual Analogue Score，VAS，Score range from 0：no pain to 10：most pain） after receiving Recombinant Human Insulin Patch ZJSRM2021

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohong X Wu, Principal Investigator — Department of Endocriology, Zhejiang Provincial People's Hospital
Locations (1):
- Zhejiang provincial people's hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
No plan to share data